CLINICAL TRIAL: NCT01081431
Title: A Multicenter, Single-arm, Open-label Phase II Study of the Safety of Lenalidomide Monotherapy and Markers for Disease Progression in Patients With IPSS Low- or Intermediate-1 Risk Myelodysplastic Syndromes (MDS) Associated With an Isolated Deletion 5q Cytogenetic Abnormality (Del 5q)
Brief Title: Safety of Lenalidomide and Markers for Disease Progression in Patients With International Prognostic Scoring System (IPSS) Low- or Intermediate-1 Risk Myelodysplastic Syndromes (MDS) With Isolated del5q
Acronym: MDS-LE-MON-5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Collaborators: ClinAssess GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MDS-PI-409; 2008-001866-10 (EudraCT Number); GMIHO-003/2008 (Other: Sponsor Code)
Record Dates: First submitted 2010-03-02; First posted 2010-03-05 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2017-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; MDS; deletion 5q; del 5q; IPSS; low risk; intermediate-1 risk; GMIHO; ClinAssess; Germing; Düsseldorf; MDS-LE-MON-5; Lenalidomide; Revlimid
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 10 mg d1-d21 of a 28-day cycle
  Other Names: CC5013; CC-5013; Revlimid

SUMMARY:
The purpose of this study is to determine the safety of lenalidomide and markers for disease progression in the treatment of IPSS low- or intermediate-1 risk MDS with isolated del5q.

DETAILED DESCRIPTION:
Lenalidomide has been successfully used in patients with MDS in several studies. A small proportion of patients with MDS and del(5q) developed leukemia while treated with Lenalidomide. Up to now it is unknown what patients are at risk to progress while being treated with Lenalidomid. Therefore it is planned to examine not only the traditional clinical parameters like disease status and proportion of blasts, but also cytogenetic findings, gene expression, antiangiogenic effect, marrow fibrosis, mesenchymal stem cell as well as mitochondrial DNA mutation at baseline and in the course of the study performed by central laboratories. Moreover, long-term data are required, e.g., with regard to the development of AML. Therefore, it is planned to collect data from all patients with MDS and del 5q (isolated, blast count <5%) in whom treatment with lenalidomide is the best therapeutic option according to the investigator's assessment in a structured fashion.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form
* Age ≥ 18 years at the time of signing the informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements
* Cytologically/histologically confirmed diagnosis of MDS with del 5q (isolated, blast count <5%), IPSS low or intermediate-1.
* Transfusion dependency with at least 1 concentrates of erythrocytes within 8 weeks prior to first administration of study drug.
* Start of treatment with lenalidomide is the best therapeutic option for the patient according to the investigator's assessment There are - apart from individual cases with erythropoetin level lower than 500 U/l and allogeneic transplantation for younger patients - no authorized alternative treatment options. Chemotherapy with low dose cytosine arabinoside may result in hematologic improvement. However, concerning the risk-benefit-assessment this chemotherapy is more unfavorable than lenalidomide due to cytopenia and mutagenic effects.
* Female subjects of childbearing potential must:

  * Understand that the study medication has a teratogenic risk
  * Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception*: (Implant,Levonorgestrel-releasing intrauterine system (IUS)**,Medroxyprogesterone acetate depot, Tubal sterilisation, Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses, Ovulation inhibitory progesterone-only pills (i.e., desogestrel))
  * Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days before the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
  * Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence

(*) Combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of VTE continues for 4 to 6 weeks after stopping combined oral contraception.

(**) Prophylactic antibiotics should be considered at the time of insertion particularly in patients with neutropenia due to risk of infection

* Male subjects must

  * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
  * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
* All subjects must

  * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
  * Agree not to share study medication with another person and to return all unused study drug to the investigator

Exclusion Criteria:

* Pregnant or lactating females
* IPSS intermediate-2 or high-risk
* Proliferative (WBC ≥ 12 x 109/L) CMML
* Any of the following laboratory abnormalities:

  * Absolute neutrophil count (ANC) < 1 x 109/L
  * Platelet count < 50 x 109/L
  * Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) > 3.0 x upper limit of normal (ULN)
  * Serum total bilirubin > 1.5 mg/dL Degree of severity of anemia is no exclusion criteria due to intensive interindividual variations of the haemoglobin value at time of transfusion.
* Prior ≥ grade-2 NCI CTCAE allergic reaction to thalidomide
* Prior desquamating (blistering) rash while taking thalidomide
* Neuropathy ≥ grade 2
* Clinically significant anemia owing to iron, B12, or folate deficiencies, or autoimmune or hereditary hemolysis or gastrointestinal bleeding (the subject must have a marrow aspirate that is evaluable for storage iron)
* Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 3 years
* Concomitant use of androgens (exception: treatment of hypogonadism)
* Concomitant use of specific treatments for MDS
* Known HIV-1 positivity
* Participation in another clinical study in the 4 weeks prior to enrollment or during this study
* Prior treatment with lenalidomide
* Any serious medical condition or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he/she participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-03-26; Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
To identify predictive factors for disease progression in patients with MDS and an isolated deletion del(5q), blast count <5%, undergoing treatment with lenalidomide | maximum 4 years

SECONDARY OUTCOMES:
Transfusion Independency on 56 consecutive days after enrollment | maximum 4 years
Cytologic Review | maximum 4 years
  Investigation of bone marrow to identify blasts, ringed sideroblasts and dysplastic changes

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Germing, Prof., Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (12):
- Germany (12):
  - Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Kath. Klinikum Duisburg, Duisburg
  - Heinrich Heine Universität Düsseldorf, Düsseldorf
  - Klinikum der J.W. Goethe Universität, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Mannheim, Mannheim
  - TU München - Klinikum rechts der Isar, München
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- See also: MDS Register — http://www.mds-register.de/